CLINICAL TRIAL: NCT00225225
Title: Rosiglitazone-Induced Weight Gain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to published data on Rosiglitazone
Sponsor: Stanford University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Marina Basina, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 96242; SPO# 34216
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

ARMS (2):
- fixed calorie (500 kcal) Reduction (Active Comparator)
  Interventions: Drug: Rosiglitazone
- Control (no diet change) (Placebo Comparator)
  Interventions: Drug: Rosiglitazone; Behavioral: dietary recommendation for weight maintenance

INTERVENTIONS:
Drug: Rosiglitazone
Behavioral: dietary recommendation for weight maintenance
  Arms: Control (no diet change)

SUMMARY:
Given the high prevalence of type 2 diabetes and the 2- to 4-fold increased risk of fatal and non-fatal coronary heart disease events in these patients, long-term glycemic control is of great importance. TZDs improves glycemic control in patients with type 2 DM as well as enhances their insulin-mediated glucose disposal. However, the improvement of glycemic control seen with TZDs may be blunted in the long run by weight gain.

Previous data on weight gain during TZD therapy in patients with type 2 DM is very sparse. It is generally assumed that an increase in adipocyte differentiation is the cause of weight gain in association with TZD treatment which may limit their use. Increased body weight assumed to compromise the positive effects of treatment. There is also a theoretical concern that, with the development of new adipocytes, future weight loss may be difficult.

However, if weight gain is primarily due to failure to adjust caloric intake in proportion to the decrease in urinary glucose loss, it is totally preventable. It has been previously shown that improvement of glycemia favored weight gain by decreasing the energy loss in the urine as glucose. Severity of weight gain appears to be proportional to the level of glycemic control achieved.

The overall goal of the proposed research is to provide the experimental evidence for the later alternative by showing that the modest weight gain that takes place in association with effective rosiglitazone treatment of hyperglycemic patients with type 2 DM is primarily due to its therapeutic efficacy. More specifically, by decreasing the caloric intake in proportion to a decrease in urinary glucose loss associated with improved glycemic control, we will be able to prevent significant weight gain following Rosiglitazone treatment. In order to provide an optimal dietary modification that can be universally applied to TZD-treated patients in clinical practice, we will have a group with a fixed amount of caloric restriction per day. It will be the first randomized controlled trial of a potential strategy for prevention of weight gain associated with thiazolidinediones.

DETAILED DESCRIPTION:
Study Design Randomized, controlled trial. Volunteers for the study will be recruited by advertisements in the local newspapers as well as through Stanford University e-mail. All studies will occur at Stanford General Clinical Research Center (GCRC).

At baseline, enrolled candidates will be required to keep a daily food and beverage record for 2 weeks as well as blood sugar log of at least 2 measurements a day (fasting and pre-dinner). Candidates will have an initial nutrition/diabetes consult with dietitian. They also will be asked to do a 24-hour urine collection once a week (2 times during the 2 week period) for quantitative assessment of glucosuria. During those 2 weeks individuals will come for GCRC outpatient visit once a week for weight, blood pressure, and blood sugar check.

After the initial two weeks, all individuals will undergo a meal profile test, after a 12-hour overnight fast, which consists of measurement of daylong plasma glucose, free fatty acids, and insulin responses to standard meals. Food for the test will be prepared by GCRC Metabolic kitchen. In order to assess the degree of postprandial and day-long hyperinsulinemia and the benefits of rosiglitazone on the metabolic abnormalities in patients with poor glycemic control, we plan to measure plasma glucose, free fatty acids, and insulin concentrations before 8 am and at hourly intervals for four hours after breakfast at 8 am and four hours after lunch at noon in response to identical test meals containing (as percentage of calories) 15% protein, 40% fat, and 45% carbohydrate. Baseline blood samples for fasting lipid and lipoprotein concentrations will be obtained after an overnight fast on the day of the meal profile. Cholesterol and lipoprotein subclasses will be analyzed by VAP-II method which is based on continuous enzymatic analysis of cholesterol and lipoprotein classes separated by a single vertical spin centrifugation using a controlled-dispersion flow analyzer. Hemoglobin A1C will be measured by an affinity chromography assay at baseline and at the end of the study.

Randomization protocol. After completion of the Meal Profile test all subjects will be started on Rosiglitazone for improvement of their glycemic control and randomized to one of the three groups (15 subjects in each group):

1. Continuation of the current diet.
2. Reduced calorie diet. Amount of reduced calories will be calculated proportionally to the calories lost via glucosuria.
3. Fixed calorie reduction diet. Reduction of daily caloric intake by 500 kcal. Rosiglitazone will be given at 4 mg for the first 4 weeks, and if tolerated, increased to 8 mg for the duration of the study. All candidates will have counseling on general meal plan with the nutritionist.

Follow-up. Subjects will be followed for 4 months. They will come to the GCRC twice a month for weight, blood pressure, blood sugar checks, and for nutrition follow-up.

End of the study measurements and clinical procedures: meal profile, lipid panel, 24-hour urine collection will be done at the end of 4 month follow-up period. Liver function tests will be done at the baseline, 4, 8, 12, and 16 weeks while on Rosiglitazone.

Outcomes: we expect to demonstrate at the end of the study that modification of the diet prevents weight gain in Rosiglitazone treated patients and to offer the optimal dietary interventions that could be applied in TZD-treated patients to minimize weight gain while effectively treating DM and insulin resistance.

Inclusion / Exclusion Inclusion criteria: 1) age between 30 and 70 years old, 2) normal chemical screening battery, 2) BMI less than 36 kg/M2, 3) non-controlled type 2 DM, defined by a fasting plasma glucose between 160 and 220 mg/dl, 4) individuals should be on a stable dose of sulfonylurea for at least one month prior to the enrollment.

Exclusion criteria: 1) liver enzymes 2.5 times above normal values, 2) chronic inflammatory, neoplastic disease, 3) subjects with clinical evidence of congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:- 1) age between 30 and 70 years old, 2) normal chemical screening battery, 2) BMI less than 36 kg/M2, 3) non-controlled type 2 DM, defined by a fasting plasma glucose between 160 and 220 mg/dl, 4) individuals should be on a stable dose of sulfonylurea for at least one month prior to the enrollment. Exclusion Criteria:- 1) liver enzymes 2.5 times above normal values, 2) chronic inflammatory, neoplastic disease, 3) subjects with clinical evidence of congestive heart failure.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-10; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
modification of the diet prevents weight gain.

SECONDARY OUTCOMES:
develop specific dietary recommendations

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Vasudevan AR, Balasubramanyam A. Thiazolidinediones: a review of their mechanisms of insulin sensitization, therapeutic potential, clinical efficacy, and tolerability. Diabetes Technol Ther. 2004 Dec;6(6):850-63. doi: 10.1089/dia.2004.6.850. PMID 15684639
- [Background] Asnani S, Richard BC, Desouza C, Fonseca V. Is weight loss possible in patients treated with thiazolidinediones? Experience with a low-calorie diet. Curr Med Res Opin. 2003;19(7):609-13. doi: 10.1185/030079903125002306. PMID 14606983
- [Background] Camp HS. Thiazolidinediones in diabetes: current status and future outlook. Curr Opin Investig Drugs. 2003 Apr;4(4):406-11. PMID 12808879
- [Background] Viberti GC. Rosiglitazone: potential beneficial impact on cardiovascular disease. Int J Clin Pract. 2003 Mar;57(2):128-34. PMID 12661797